CLINICAL TRIAL: NCT07268781
Title: The Effect of Golden Rice Cookies With Piper Crocatum Extract on Lipid Profile Control in Patients With Diabetes Mellitus
Brief Title: Impact of Golden Rice-Piper Crocatum Cookies on Lipid Control in Diabetes Mellitus Patients
Acronym: GRPC-DM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Altje Suwardi Abram, S.Kep.,Ns, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UH2507094
Record Dates: First submitted 2025-09-30; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus (DM); Dyslipidemia; Lipid Profile; Functional Food; Nutritional Intervention; Cardiovascular Risk Factor
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: This study is an interventional clinical trial with a parallel-group design to evaluate the effect of Golden Rice cookies enriched with Piper crocatum extract on lipid profile control in patients with Type 2 Diabetes Mellitus. Participants will be divided into two groups: the intervention group, which will receive Golden Rice cookies containing Piper crocatum extract for 28 consecutive days, and the control group, which will receive standard care (placebo) without the functional food intervention. The study follows a pre-test and post-test control group design, where lipid profile parameters including total cholesterol, LDL, HDL, and triglycerides will be assessed at baseline and after the 28-day intervention period. The allocation is randomized, while masking is not applied due to the nature of the dietary intervention. The primary purpose of this study is treatment, aiming to improve lipid metabolism, reduce dyslipidemia, and prevent cardiovascular complications in patients with
Who Masked: Participant
Masking Description: Participants will not be informed about whether they are in the intervention or control group, since both groups will receive packaged cookies that appear identical. Investigators and care providers will know the allocation in order to ensure proper delivery of the intervention, but outcome assessors and laboratory personnel measuring lipid profiles will remain blinded to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golden Rice cookies With Piper Crocatum extract (Experimental): Participants will receive Golden Rice cookies enriched with Piper crocatum extract as a daily dietary supplement for 28 consecutive days. The cookies are formulated as a functional food, providing β-carotene from Golden Rice and polyphenols from Piper crocatum, which have antioxidant, anti-inflammatory, and lipid-modulating properties. The intervention aims to improve lipid metabolism by reducing total cholesterol, LDL, and triglycerides while increasing HDL levels in patients with Diabetes Mellitus.
  Interventions: Dietary Supplement: Golden Rice cookies with Piper crocatum Extract
- Active Comparator (Control) (Active Comparator): Participants will receive Golden Rice cookies without Piper crocatum extract, identical in appearance and packaging to the intervention cookies, for 28 consecutive days. This control is designed to maintain participant blinding and to serve as a comparison for evaluating the specific effects of Piper crocatum extract on lipid profile outcomes.
  Interventions: Dietary Supplement: Placebo Cookies (Control)

INTERVENTIONS:
Dietary Supplement: Golden Rice cookies with Piper crocatum Extract — Golden Rice cookies enriched with Piper crocatum extract, formulated as a functional food containing β-carotene and polyphenols with antioxidant, anti-inflammatory, and lipid-modulating properties. Participants will consume the cookies daily for 28 consecutive days in addition to their standard diabetes management. This intervention is designed to improve lipid metabolism and reduce dyslipidemia in patients with Diabetes Mellitus.
  Arms: Golden Rice cookies With Piper Crocatum extract
Dietary Supplement: Placebo Cookies (Control) — Placebo cookies without Golden Rice or Piper crocatum extract, identical in appearance, taste, and packaging to the intervention cookies. Participants will consume placebo cookies daily for 28 consecutive days along with their standard diabetes management. This placebo is used to maintain participant blinding and provide a valid comparison.
  Arms: Active Comparator (Control)

SUMMARY:
People with diabetes often experience abnormal blood fat levels, known as dyslipidemia, which increase the risk of heart disease and stroke. The aim of the study, researchers are exploring a natural and practical solution through a healthy snack in the form of cookies. These cookies are made from Golden Rice, which is rich in beta-carotene as a natural antioxidant, and Piper crocatum (red betel leaf) extract, which contains polyphenols and flavonoids that may help lower cholesterol, reduce inflammation, and protect blood vessels. In this study, patients with diabetes will consume the cookies for 28 days, and their blood fat levels will be measured before and after the intervention. The results will then be compared with those of a control group who receive the Golden rice cookies without piper crocatum extract. This research aims to show that Golden Rice with Piper crocatum extract cookies can reduce bad cholesterol and triglycerides, increase good cholesterol, and serve as a safe, affordable, and acceptable food option to support daily diabetes care. If successful, this approach may offer patients and families a simple way to help prevent complications and improve quality of life, alongside regular treatment and lifestyle changes.

DETAILED DESCRIPTION:
This clinical trial evaluates the effect of Golden Rice cookies enriched with Piper crocatum (red betel leaf) extract on lipid profile control in patients with type 2 diabetes mellitus. The intervention is designed as a short-term, food-based strategy to complement existing diabetes management by integrating functional food into daily dietary practice.

The rationale for this approach is based on evidence that beta-carotene from Golden Rice and polyphenols from Piper crocatum exert antioxidant, anti-inflammatory, and lipid-lowering activities. Combining these bioactive compounds in the form of cookies provides a culturally acceptable, affordable, and practical dietary intervention. The cookie format was selected due to its high acceptance, ease of distribution, and potential to improve adherence compared with capsule or extract preparations.

This trial uses a controlled pre-post design to compare changes in lipid biomarkers between the intervention and control groups over 28 days. Key outcomes include serum levels of LDL cholesterol, HDL cholesterol, triglycerides, and total cholesterol. The study also explores potential synergistic effects on oxidative stress and inflammatory processes associated with dyslipidemia in diabetes.

By translating the concept of functional food into a practical dietary item, this study aims to generate evidence for its role as an adjunctive therapy in diabetes care. Findings are expected to inform future dietary guidelines and nursing interventions, particularly in community-based settings where accessibility, patient adherence, and cost-effectiveness are critical considerations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-59 years.
* Patients diagnosed with Type 2 Diabetes Mellitus based on medical records at Tambu Primary Health Center.
* Able to read and communicate effectively with healthcare staff.
* Permanent resident in the Tambu area.
* Willing to participate in the intervention and follow-up evaluations for the duration of the study.

Exclusion Criteria:

* Pregnant or breastfeeding women, or those currently undergoing a pregnancy program.
* Patients with mental health disorders.
* Patients with severe comorbidities affecting lipid metabolism, such as chronic kidney disease (CKD), hepatitis, congestive heart failure, stroke, or acute coronary syndrome within the past 3 months.
* Patients who have consumed herbal supplements or high-dose antioxidants within the last month.
* Patients with severe gastrointestinal disorders, such as chronic diarrhea.
* Patients with a history of allergy to any ingredients used in the study intervention.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total Cholesterol (mg/dL) | Baseline (Day 0) and after 28 days of intervention
  Serum total cholesterol will be measured to assess the effect of Golden Rice cookies enriched with Piper crocatum extract on lipid control in patients with diabetes mellitus.
Change in Low-Density Lipoprotein (LDL) Cholesterol (mg/dL) | Baseline (Day 0) to Day 28
  LDL cholesterol levels will be measured to evaluate changes following the 28-day intervention
Change in High-Density Lipoprotein (HDL) Cholesterol (mg/dL) | Baseline (Day 0) to Day 28
  HDL cholesterol levels will be measured to determine improvement in protective lipid fractions.
Change in Triglycerides (mg/dL) | Baseline (Day 0) to Day 28
  Serum triglyceride levels will be measured to assess metabolic lipid response to the intervention.

SECONDARY OUTCOMES:
Participant adherence Rate (%) | Baseline to Day 28
  Daily adherence to the assigned cookie regimen will be monitored using participant self-report checklists and confirmed by the count of returned empty packaging during weekly follow-up visits. Adherence will be reported as the percentage of prescribed doses consumed over the 28-day intervention.
Incidence of Adverse Events (Number of Participants) | Baseline to Day 28
  All adverse events and signs of intolerance (e.g., gastrointestinal symptoms, allergic reactions) potentially associated with the intervention will be documented throughout the study period. Events will be classified by type, severity, onset, duration, and relationship to the study product. Results will be reported as the number and percentage of participants experiencing at least one adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: ANDINA SETYAWATI, PhD, S.Kep., Ns., M.Kep., Study Director — Hasanuddin University, Faculty of Nursing
Locations (2):
- Indonesia (2):
  - Tambu Primary Health Center (Puskesmas Tambu), Donggala, Central Sulawesi
  - RSUD Anutapura Palu, Palu, Central Sulawesi

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) for this study.

REFERENCES:
- [Background] Setyawati A, Saleh A, Tahir T, Yusuf S, Syahrul S, Aminuddin A, Raihan M, Jafar N, Hamzah H, Arfian N. Matrix Metalloproteinase-9 Testing of Golden Rice Cookies With Piper Crocatum Active Extract for Preventing Foot Ulcers in Patients With Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 29;13:e49940. doi: 10.2196/49940. PMID 38422498
- [Result] https://jppres.com/jppres/pdf/vol13/jppres25.2499_13.6.1847.pdf
- [Result] Setyawati A, Wahyuningsih MSH, Nugrahaningsih DAA, Effendy C, Fneish F, Fortwengel G. Piper crocatum Ruiz & Pav. ameliorates wound healing through p53, E-cadherin and SOD1 pathways on wounded hyperglycemia fibroblasts. Saudi J Biol Sci. 2021 Dec;28(12):7257-7268. doi: 10.1016/j.sjbs.2021.08.039. Epub 2021 Aug 19. PMID 34867030
- See also: Official website of the Faculty of Nursing, Universitas Hasanuddin. — https://nursing.unhas.ac.id/
- See also: Universitas Hasanuddin official website. — https://unhas.ac.id/